CLINICAL TRIAL: NCT05422326
Title: A Phase 2, Randomized, Study to Evaluate Safety and Immunogenicity of One or Two Heterologous Booster Vaccinations With an MF59-adjuvanted, Cell Culture-derived H5N6 Influenza Vaccine in Adults Primed With MF59-adjuvanted, Cell Culture-derived H5N1 Influenza Vaccine or Unprimed
Brief Title: A Study to Evaluate Safety and Immunogenicity of One or Two Booster Vaccinations With H5N6 Influenza Vaccine in Adults Primed With H5N1 Influenza Vaccine or Unprimed
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seqirus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V89_18E1
Record Dates: First submitted 2022-06-14; First posted 2022-06-16 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Influenza, Human; Influenza in Birds; Respiratory Tract Infections; Infections; Orthomyxoviridae Infections; RNA Virus Infections; Virus Diseases; Respiratory Tract Diseases
Keywords: Influenza; Pandemic; Vaccine; H5N1; H5N6; Flu; MF59; Avian
MeSH Terms: conditions — Influenza, Human; Influenza in Birds; Respiratory Tract Infections; Infections; Orthomyxoviridae Infections; RNA Virus Infections; Virus Diseases; Respiratory Tract Diseases

STUDY DESIGN:
Intervention Model Description: Eligible subjects, who received 2 doses of aH5N1c in the parent study V89_18 are randomized in a 1:1 ratio to group 1 (two aH5N6c vaccinations, 3 weeks apart) or group 2 (aH5N6c vaccination and placebo, 3 weeks apart).
  Eligible subjects, who received placebo in the parent study are allocated to group 3 (two aH5N6c vaccinations, 3 weeks apart).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Experimental): Eligible subjects who received 2 doses of aH5N1c in the parent study V89_18 and have been randomized to receive two aH5N6c vaccinations, 3 weeks apart
  Interventions: Biological: aH5N6c on Day 1; Biological: aH5N6c on Day 22
- Group 2 (Experimental): Eligible subjects who received 2 doses of aH5N1c in the parent study V89_18 and have been randomized to receive an aH5N6c vaccination on Day 1 and saline placebo on Day 22
  Interventions: Biological: aH5N6c on Day 1; Biological: Placebo on Day 22
- Group 3 (Experimental): Eligible subjects who received placebo in the parent study V89_18 receive two aH5N6c vaccinations, 3 weeks apart.
  Interventions: Biological: aH5N6c on Day 1; Biological: aH5N6c on Day 22

INTERVENTIONS:
Biological: aH5N6c on Day 1 — MF59-adjuvanted cell-culture derived subunit inactivated monovalent A/H5N6 vaccine (aH5N6c) for intramuscular (IM) administration, containing 7.5 μg H5N6 hemagglutinin (HA) (A/Guangdong/18SF020/2018 (H5N6)-like) + 0.25 mL MF59 (approximately 0.5 mL total volume)
Biological: aH5N6c on Day 22 — MF59-adjuvanted cell-culture derived subunit inactivated monovalent A/H5N6 vaccine (aH5N6c) for intramuscular (IM) administration, containing 7.5 μg H5N6 HA (A/Guangdong/18SF020/2018 (H5N6)-like) + 0.25 mL MF59 (approximately 0.5 mL total volume) given 3 weeks after the first aH5N6c vaccination
  Arms: Group 1; Group 3
Biological: Placebo on Day 22 — Saline placebo (sterile, 0.5 mL) given 3 weeks after the aH5N6c vaccination
  Arms: Group 2

SUMMARY:
This is a Phase 2, randomized, multi-center study in approximately 300 adults who received 2 doses of aH5N1c or placebo in and completed the parent study V89_18 in the <65 years of age cohort. The study investigates whether two priming doses of MF59-adjuvanted H5N1 cell culture-derived vaccine (aH5N1c) followed by one or two booster vaccinations with a MF59-adjuvanted H5N6 cell culture derived vaccine (aH5N6c) 3 weeks apart elicit immune responses to the antigens used for priming (H5N1) and boosting (H5N6) after first and second heterologous booster vaccination.

Eligible subjects, who received 2 doses of aH5N1c in the parent study V89_18 are randomized in a 1:1 ratio to receive either two aH5N6c vaccinations, 3 weeks apart (group 1) or an aH5N6c vaccination on Day 1 and saline placebo on Day 22 (group 2). Eligible subjects, who received placebo in the parent study will receive two aH5N6c vaccinations, 3 weeks apart (group 3). After the second vaccine administration, subjects are monitored for approximately 6 months for safety and antibody persistence. The total study duration will be approximately 7 months per subject.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who received 2 doses of aH5N1c vaccine or placebo in and completed the parent study V89_18 in the <65 years of age cohort.
* Individuals who can comply with study procedures including follow-up.

Exclusion Criteria:

* Females of childbearing potential who are pregnant, lactating, or who have not adhered to a specified set of contraceptive methods from at least 30 days prior to study entry and who do not plan to do so until at least 30 days after the last study vaccination.
* Progressive, unstable or uncontrolled clinical conditions.
* Hypersensitivity, including allergy, to any component of vaccines, medicinal products or medical equipment whose use is foreseen in this study.
* Clinical conditions representing a contraindication to intramuscular vaccination and blood draws.
* Abnormal function of the immune system.
* History of any medical condition considered an adverse event of special interest (AESI).
* Received immunoglobulins with immunomodulating effects or any blood products within 180 days prior to informed consent.
* Subjects, who received an influenza H5 vaccine other than in the V89_18 parent study or have a history of H5 influenza infection prior to enrollment.
* Received an investigational or non-registered medicinal product within 30 days prior to informed consent.
* Individuals who received any other vaccines [except corona virus disease 2019 (COVID-19) vaccines] within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to enrollment in this study or who are planning to receive any vaccine within 28 days from the study vaccination.
* Receipt of any COVID-19 vaccine within 7 days prior to enrollment or plan to receive any COVID-19 vaccine within 7 days from study vaccination.
* Acute (severe) febrile illness.
* A known history of Guillain-Barre Syndrome or other demyelinating diseases such as encephalomyelitis and transverse myelitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2023-03-24 (Actual)

PRIMARY OUTCOMES:
Geometric Mean Titer (GMT) of hemagglutination inhibition (HI) antibodies against H5N6 strain | Day 1, Day 8, Day 22, Day 43
  GMT pre-vaccination, 1 and 3 weeks post-vaccination 1, and 3 weeks post-vaccination 2
Geometric Mean Fold Increase (GMFI) of HI antibodies against H5N6 strain | Day 1, Day 8, Day 22, Day 43
  GMFI 1 and 3 weeks post-vaccination 1, and 3 weeks post-vaccination 2 compared to pre-vaccination (Day 1)
Percentage of subjects with HI titers ≥1:40 against H5N6 strain | Day 1, Day 8, Day 22, Day 43
  Pre-vaccination, 1 and 3 weeks post-vaccination 1, and 3 weeks post-vaccination 2
Percentage of subjects with seroconversion against H5N6 strain | Day 8, Day 22, Day 43
  Seroconversion 1 and 3 weeks post-vaccination 1, and 3 weeks post-vaccination 2, defined as a ≥4-fold increase in HI titer post-vaccination in those with pre-vaccination titer ≥1:10, or a post-vaccination HI titer ≥1:40 for subjects with baseline titer <1:10

SECONDARY OUTCOMES:
GMT of HI antibodies against H5N1 strain | Day 1, Day 8, Day 22, Day 43, Day 202
  GMT pre-vaccination, 1 and 3 weeks post-vaccination 1, and 3 weeks and 6 months post-vaccination 2
GMFI of HI antibodies against H5N1 strain | Day 1, Day 8, Day 22, Day 43, Day 202
  GMFI 1 and 3 weeks post-vaccination 1, and 3 weeks and 6 months post-vaccination 2 compared to pre-vaccination (Day 1)
Percentage of subjects with HI titers ≥1:40 against H5N1 strain | Day 1, Day 8, Day 22, Day 43, Day 202
  Pre-vaccination, 1 and 3 weeks post-vaccination 1, and 3 weeks and 6 months post-vaccination 2
Percentage of subjects with seroconversion against H5N1 strain | Day 8, Day 22, Day 43, Day 202
  Seroconversion 1 and 3 weeks post-vaccination 1, and 3 weeks and 6 months post-vaccination 2, defined as a ≥4-fold increase in HI titer post-vaccination in those with pre-vaccination titer ≥1:10, or a post-vaccination HI titer ≥1:40 for subjects with baseline titer <1:10
GMT of HI antibodies against H5N6 strain | Day 202
  GMT 6 months post-vaccination 2
GMFI of HI antibodies against H5N6 strain | Day 1, Day 202
  GMFI 6 months post-vaccination 2 compared to pre-vaccination (Day 1)
Percentage of subjects with HI titers ≥1:40 against H5N6 strain | Day 202
  6 months post-vaccination 2
Percentage of subjects with seroconversion against H5N6 strain | Day 202
  Seroconversion 6 months post-vaccination 2, defined as a ≥4-fold increase in HI titer post-vaccination in those with pre-vaccination titer ≥1:10, or a post-vaccination HI titer ≥1:40 for subjects with baseline titer <1:10
Frequency and severity of solicited local and systemic adverse events (AEs) | Day 1 through Day 7 and Day 22 through Day 28
  For 7 days following each vaccination
Frequency and severity of unsolicited AEs | Day 1 through Day 43
  For 3 weeks following each vaccination
Frequency and severity of serious AEs (SAEs), AEs leading to withdrawal, AEs of special interest (AESI) and medically attended AEs (MAAEs) | Day 1 through Day 202
  From vaccination until study completion

CONTACTS AND LOCATIONS:
Overall Officials: Therapeutic Area Head, Study Chair — Seqirus
Locations (18):
- United States (18):
  - Optimal Research, LLC, Huntsville, Alabama
  - Clinical Research Consortium Arizona, Tempe, Arizona
  - California Research Foundation, San Diego, California
  - Clinical Research Consulting, LLC, Milford, Connecticut
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - Optimal Research, LLC, Melbourne, Florida
  - Great Lakes Clinical Trials LLC, Chicago, Illinois
  - Heartland Research Associates, LLC, Wichita, Kansas
  - The Center for Pharmaceutical Research, Kansas City, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Rochester Clinical Research, Inc, Rochester, New York
  - PMG Research of Raleigh, Raleigh, North Carolina
  - AccellaCare, Winston-Salem, North Carolina
  - Aventiv Research, Columbus, Ohio
  - Biogenics Research Institute, San Antonio, Texas
  - J. Lewis Research, Inc/Foothill Family Clinic North, Salt Lake City, Utah
  - J. Lewis Research, Inc/Foothill Family Clinic South, Salt Lake City, Utah
  - J. Lewis Research, Inc/Jordan River Family Medicine, South Jordan, Utah

IPD SHARING:
Plan to Share IPD: Undecided